CLINICAL TRIAL: NCT05182671
Title: Relationship Between Pelvic Angle, Femoral Anteversion, and Hip Muscle Strength Ratios in Children With Bladder-bowel Dysfunction
Brief Title: Relationship Between Pelvic Angle, Femoral Anteversion, and Hip Muscle Strength Ratios in Bladder-bowel Dysfunction
Status: Completed | Type: Observational
Sponsor: Halil Tugtepe (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor-Investigator, Halil Tugtepe, Professor, Dr. (MD), Tugtepe Pediatric Urology Clinic
Organization: Tugtepe Pediatric Urology Clinic (Other)
Other Study IDs: TUGTEPEPUC
Record Dates: First submitted 2021-11-21; First posted 2022-01-10 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Bladder and Bowel Dysfunction, Femoral Anteversion; Bladder and Bowel Dysfunction, Hip Strength Ratios; Bladder and Bowel Dysfunction, Pelvic Angle
MeSH Terms: conditions — Intestinal Diseases | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children diagnosed with bowel and bladder dysfunction: Children who are between the ages of 5-12 and diagnosed with bladder- bowel dysfunction by pediatric urologist.
  Interventions: Other: Scales and measurements for bladder and bowel dysfunction, pelvic angle, proximal hip strength, femoral hip anteversion

INTERVENTIONS:
Other: Scales and measurements for bladder and bowel dysfunction, pelvic angle, proximal hip strength, femoral hip anteversion — Assessments Children whose physical examination has been completed and diagnosed with BBD will be evaluated with following assessments.
  Demographic Data Form Questionnaire Forms Dysfunctional Voiding and Incontinence Scoring System Bladder Diary Bowel Diary EMG-uroflowmetry Ultrasonography
  Post Voiding Residual Measurement:
  Bladder wall thickness
  Pelvic Floor Muscle Activation Measurement:
  Pelvic Floor Muscle Strength Assessment:
  Hip agonist-antagonist muscle ratios Pelvic angle measurement Femoral anteversiyon angle measurement
  Femoral internal and external rotation angle:

SUMMARY:
Bladder and bowel dysfunction is a combination of lower urinary tract and bowel dysfunction seen in children over 5 years of age without identifiable or discernible neurological abnormalities. The proper functioning of the bladder, bowel, nerves, pelvic floor muscles and related anatomical structures provides the bowel and lower urinary tract function. Dysfunction of any structure of the pelvic floor can potentially cause to bladder and bowel dysfunction. The ability of the pelvic floor muscles to perform the correct contraction and relaxation function is also closely related to the position of the pelvis, muscle strength of the hip muscles, and femoral anteversion. Disruption of one of the links forming the chain causes a change in the mobility and stability of all mechanically related structures and may affect the optimal force that the pelvic floor muscles can produce.

As far as investigators know, there is no study in the literature examining the relationship between BBD and pelvic angle, femoral anteversion angle, femoral internal/external rotation angle ratio and hip muscle strength ratios in children with bladder-bowel dysfunction. Considering the close relationship between pelvis position, hip muscle strength, and femoral anteversion with the pelvic floor, investigators think that this relationship should be evaluated in children with BBD and will contribute to the literature.

DETAILED DESCRIPTION:
Bladder and bowel dysfunction (BBD) is a combination of lower urinary tract (LUT) and bowel dysfunction seen in children over 5 years of age without identifiable or discernible neurological abnormalities. Constipation and fecal incontinence are common bowel dysfunctions. Common lower urinary tract dysfunction (LUTD) symptoms of BBD include dysuria, urgency, urinary frequency, difficulty in initiating urine, daytime incontinence, enuresis, straining, delayed voiding, and urinary retention. Urological conditions such as overactive bladder, underactive bladder and dysfunctional voiding can also be part of BBD.

The proper functioning of the bladder, bowel, nerves, pelvic floor muscles and related anatomical structures provides the bowel and LUT function. The pelvic floor is a structure located at the base of the pelvis, consisting of smooth and striated muscle sphincters, endopelvic fascia, connective tissue and ligaments, mucosal and vascular tissues, levator ani and more superficial perineal muscles. It actively supports the pelvic organs (bladder, bowel, uterus) and provides continence. Dysfunction of any structure of the pelvic floor can potentially cause to bladder and bowel dysfunction.

The ability of the pelvic floor muscles to perform the correct contraction and relaxation function is also closely related to the position of the pelvis, muscle strength of the hip muscles, and femoral anteversion. The pelvis and lower extremity consist of interconnected closed chain structures. The movement of any link in the chain depends on the movement of the other links. For this reason, disruption of one of the links forming the chain causes a change in the mobility and stability of all mechanically related structures and may affect the optimal force that the pelvic floor muscles can produce.

As far as investigators know, there is no study in the literature examining the relationship between BBD and pelvic angle, femoral anteversion angle, femoral internal/external rotation angle ratio and hip muscle strength ratios in children with bladder-bowel dysfunction. Considering the close relationship between pelvis position, hip muscle strength, and femoral anteversion with the pelvic floor, investigators think that this relationship should be evaluated in children with BBD and will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 5-12
* To be diagnosed with bladder- bowel dysfunction

Exclusion Criteria:

* To be younger than 5 years old
* To have an orthopedic disease that would prevent the evaluation
* To have anatomical changes in the urinary system
* To have having a neurological disorder
* To have cognitive impairment and mental retardation
* To have an orthopedic surgery that can change pelvis and lower extremity biomechanics

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who are between 5-12 years old, diagnosed with bladder bowel dysfunction.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Femoral anteversion angle measurement | Baseline
  Hip anteversion was measured using the Craig test with the subject in the prone position and the knee flexed to 90°. The examiner passively rotates the hip, palpating the trochanter major, until the most prominent part of the trochanter reaches its most lateral position. The angle between the true vertical and the shaft of the tibia was measured to the nearest degree, using a Accurate Compass smartphone inclinometer.
Pelvic angle measurement | Baseline
  The inferior prominence of the anterior superior iliac spine (ASIS) and the most prominent aspect of the posterior superior iliac spine (PSIS) were identified with palpation, and pelvic angle was measured as the angle formed between the horizontal plane and a line from ASIS and PSIS landmarks using an inclinometer (Performance Attainment Associates, St Paul, MN). A positive value reflected an anterior pelvic tilt (ASIS sitting lower than the PSIS).
Hip agonist-antagonist muscle ratios | Baseline
  In the isometric muscle strength measurement procedure, each test position was evaluated with 2 repetitions of submaximal force for familiarization and 3 evaluations were taken with maximal force. Each test lasted 5 seconds, with 30-second breaks between trials. A 1-minute break was given between different measurements. MicroFET(Draper, UT) hand dynamometer was used for muscle strength measurement. The order of strength testing was randomized. The dynamometer is fixed to the leg with the help of a strap. Force values are measured in kilograms and normalized to body mass using the following formula:(kg power/kg body mass)x100. The intrarater reliability study will be completed before participants' measurements begin to be taken. Hip abductor, adductor, flexor, extensor, internal rotation, external rotation muscle strength is measured. Hip adductor/abductor, medial/lateral rotator, and flexor/extensor strength ratios muscle strength ratios will be evaluated.

SECONDARY OUTCOMES:
Dysfunctional Voiding and Incontinence Scoring System | Baseline
  Dysfunctional Voiding and Incontinence Scoring System (DVISS) is a 13-item questionnaire. Parents are the target audience. DVISS scores are based on the estimated odds ratio for each question between cases and controls. For example, 1 point is awarded if the odds ratio value is between 2 and 10, and 5 points if it is greater than 50. The total score can range from 0 to 35. A cut-off value of 8.5 shows 90% specificity and sensitivity in detecting BBD.
EMG-uroflowmetry | Baseline
  In the uroflowmetry evaluation, when the patient's urge to urinate occurs, urination will be requested into the AYMED® brand EMG uroflowmetry pot with a sensor system. Stool support will be provided to ensure suitable toilet position in children whose feet do not touch the ground during the test measurement. In order to minimize the external factors that will affect the voiding pattern, there will be no one other than the patient in the uroflowmetry room. The parameters obtained as a result of the measurement will enable us to interpret the bladder's emptying phase.
Ultrasonography - Post Voiding Residual Measurement, Bladder thickness | Baseline
  Telemed® brand transabdominal ultrasound device will be used, and measurements will be made from the suprapubic region. During the measurement, the patient will be positioned in the supine position and the knees will be slightly flexed and supported with a towel under the knee. The volume values in mm3 calculated by the probe in the coronal and sagittal regions will be automatically multiplied by the ultrasound system and the residual urine remaining in the bladder will be calculated in cc. The standard method should be used for pelvic voiding residual measurements.
Pelvic Floor Muscle Activation Measurement: | Baseline
  The pelvic floor physiotherapist positions the participant in the butterfly position with support under the legs while lying on their back. Before EMG evaluation, all participants are taught to perform isolated contraction and relaxation of the pelvic floor muscles without the use of accessory muscles by anus palpation. Two superficial electrodes (30 mm diameter (VS30)) are then placed bilaterally adjacent to the mucocutaneous line of the anus at 2 and 7 o'clock to prevent cross-talking (electrodes interference and artifact formation). The reference surface electrode is placed on the inside of the right thigh.
  After proper placement of the electrodes, pelvic floor muscle activity will be measured with the NeuroTrac Myoplus4 Pro device.
Pelvic Floor Muscle Strength Assessment: | Baseline
  Manual muscle testing is a subjective assessment method. First, the child is taught to contract the pelvic floor muscles in the litotomy position (supine, butterfly position). The therapist places the index finger on the anus (perceiving contraction of the external anal sphincter), asking child's to contract the pelvic floor muscles as if she were holding child's stool or urine. The therapist then asks the child to contract the pelvic floor muscles as the muscles teach the correct contraction.
  With the manual muscle test, the strength, fatigue time and endurance of the pelvic floor muscles are evaluated. Evaluation of pelvic floor muscles in children is evaluated by palpation over the external anal sphincter, and the following grading method is used.
  Modified Oxford Scale 0= no contraction
  1= vibration 2 = weak contraction 2+= contraction without movement 3 = contraction with movement 3+= strong contraction
Femoral internal and external rotation angle | Baseline
  Passive hip internal rotation and external rotation were measured with a standard goniometer, with the child lying face down on the table in the prone position. The thigh was carefully positioned to 0° hip abduction or adduction and the contralateral leg to approximately 20° abduction. Pelvis is stabilized by another physiotherapist and examiner measured range of motion by bringing the leg to a firm end point of both IR and ER. The measurement was made by passively bringing the leg to its end point in both internal and external rotation, without lifting the pelvis from the ground. Angle measurement will be made with Accurate Compass smartphone inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Aygül Köseoğlu, PT, MSc, Principal Investigator — Tuğtepe Pediatric Urology Clinic; Halil Tuğtepe, MD, Prof Dr,, Study Chair — Tuğtepe Pediatric Urology Clinic; Pelin Pişirici, PT, PhD, Study Director — Bahçeşehir University Faculty of Health Sciences; Tuğçe Atalay, PT, Study Chair — Tuğtepe Pediatric Urology Clinic; Ece Zeynep Saatçi, PT, Study Chair — Tuğtepe Pediatric Urology Clinic; Melis Ünal, PT, Study Chair — Tuğtepe Pediatric Urology Clinic
Locations (1):
- Private Tugtepe Pediatric Urology Clinic, Istanbul, Turkey (Türkiye)